CLINICAL TRIAL: NCT06432361
Title: Resource Allocation for Alcohol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jennifer Cadigan, Assistant Professor, Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00018018; 1R34AA029478-01A1 (NIH)
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resource Allocation Intervention (Experimental): Participants will complete a 3 week monitoring period of daily surveys assessing time spent in various domains during the time, alcohol use, personal goals, and money spent on alcohol and substance-free activities. Each daily survey should take no longer than 5 minutes to complete.
  Those in the intervention condition will receive weekly personalized information summarizing the previous week's resource allocation (e.g., personalized information on how they spent their time and money) in relation to their personal goals, interests, and alcohol use. They will also see a summary of how they spent their time and money in relation to their set goals for the week. The information in the intervention feedback will be obtained from participant's responses to the daily surveys on how they spent their time and money each day. Reviewing the intervention feedback should take no longer than 10 minutes.
  Interventions: Behavioral: Resource Allocation
- Assessment only control (Active Comparator): Participants will complete a 3 week monitoring period of daily surveys assessing time spent in various domains during the time, alcohol use, personal goals, and money spent on alcohol and substance-free activities. Each daily survey should take no longer than 5 minutes to complete.
  Interventions: Other: assessment only control

INTERVENTIONS:
Behavioral: Resource Allocation — Those in the intervention condition will receive weekly personalized information summarizing the previous week's resource allocation (e.g., personalized information on how they spent their time and money) in relation to their personal goals, interests, and alcohol use. They will also see a summary of how they spent their time and money in relation to their set goals for the week The information in the intervention feedback will be obtained from participant's responses to the daily surveys on how they spent their time and money each day. Reviewing the intervention feedback should take no longer than 10 minutes.
  Arms: Resource Allocation Intervention
Other: assessment only control — participants will complete a 3 week monitoring period of daily surveys assessing time spent in various domains during the time, alcohol use, personal goals, and money spent on alcohol and substance-free activities. Each daily survey should take no longer than 5 minutes to complete.
  Arms: Assessment only control

SUMMARY:
A total of 150 young adults (ages 21-29) will be randomized to receive a brief alcohol intervention (intended to reduce alcohol-related resource allocation (e.g., time and money spent on alcohol), alcohol consumption, and alcohol related consequences) or an assessment only control condition.

All participants will complete a 3 week monitoring period of daily surveys assessing time spent in various domains, alcohol use, personal goals, and money spent on alcohol and substance-free activities. Those in the intervention condition will receive weekly personalized information summarizing the previous week's resource allocation.

All participants will complete a 1 and 3 month follow up survey. Participants can earn up to $126 for completing all study components.

ELIGIBILITY:
Inclusion Criteria:

* 1)21-29 years old, 2) reside within WA state, 3) report drinking 2+ days per week, on average, in the last six months, 4) report 4+ heavy drinking episodes (4+/5+ for women/men) in the past month,

Exclusion Criteria:

* 1) currently enrolled in a 4-year college, 2) currently in or seeking treatment for alcohol use

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Standard drinks containing alcohol- | past 1 month
  We will assess the number of standard drinks, containing alcohol in a typical week collected on the Daily Drinking Questionnaire DDQ; Collins et al., 1985; Kivlahan et al., 1990)
Alcohol-related problems | past 1 month
  We will assess the number of alcohol-related consequences experienced using the Rutgers Alcohol Problem Index.
Alcohol Demand | past 1 month
  Alcohol demand will be assessed with the Alcohol Purchase Task.
Time allocation | past 1 month
  Time allocation will be assessed (Murphy et al.,2012) where participants will indicate, on average, how many hours they spend in a typical week in various domains including alcohol-related domains.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Cadigan, PhD, Principal Investigator — University of Washington